CLINICAL TRIAL: NCT04313361
Title: China Observational Study of Smoking Cessation Patterns in Patients Undergoing Lung Surgery (CHAMPION Study)
Brief Title: A Study of Smoking Cessation Patterns in Participants Undergoing Lung Surgery
Acronym: CHAMPION
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson (China) Investment Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108767; NOPRODLUC4001 (Other: Johnson & Johnson (China) Investment Ltd.)
Record Dates: First submitted 2020-03-05; First posted 2020-03-18 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Lung Neoplasms; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Lung Neoplasms; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Smokers or Recent Smoking Quitters who Have lung Surgery: The enrolled eligible participants, that is smokers or recent smoking quitters, will be assessed for the current smoking status and smoking cessation attempts during the perioperative period, to describe postoperative complications (PCs) including postoperative pulmonary complications (PPCs) following a lung surgery, and to describe the smoking cessation methods and services participants received from their health care professionals (HCPs) and participant's satisfaction among participants with lung cancer, chronic obstructive pulmonary disorder (COPD), a pulmonary lesion (example nodule, ground glass opacity) or other pulmonary conditions who are admitted to the thoracic surgical unit of the participating hospitals in China.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No drug will be administered as part of this study.

SUMMARY:
The purpose of this study is to assess the current smoking status and smoking cessation attempts among smokers or recent smoking quitters during the perioperative period, to describe postoperative pulmonary complications (PPCs) and other postoperative complications (PCs) following a lung surgery, and to describe the smoking cessation methods and services patients received from their health care professionals (HCPs) and participant's satisfaction among participants with lung cancer, chronic obstructive pulmonary disorder (COPD), a pulmonary lesion (example, nodule, or ground glass opacity) or other pulmonary conditions who are admitted to the thoracic surgical unit of the participating hospitals in China.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have been scheduled for an elective lung surgery by the treating physician's judgement, due to the following conditions: known lung cancer, COPD, a pulmonary lesion (example. nodule, ground glass opacity) or other pulmonary conditions
* Smokers who are or were smoking on average no fewer than 5 cigarettes per day for equal or more than 3 years within 3 months prior to the scheduled surgery, or recent smoking quitters with a history of smoking on average no fewer than 5 cigarettes per day for equal or more than 3 years, who quit smoking between 3 months and 5 years prior to the scheduled surgery
* Being willing to participate the study and sign the participant informed consent form (ICF)

Exclusion Criteria:

* Participants who have emergency lung surgery due to accident or injury
* Participants are not likely to be able to complete the 6-month follow-up after the lung surgery

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult participant with lung cancer, chronic obstructive pulmonary disorder (COPD), a pulmonary lesion, or other pulmonary conditions with a scheduled lung surgery and their treating health care providers (HCPs) from three participating hospitals in China.
Sampling Method: Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Smokers and Recent Smoking Quitters at Baseline Prior to the Surgery | Baseline Prior to the Surgery
  Percentage of smokers and recent smoking quitters at baseline prior to the surgery will be reported.
Smoking Dependence Among Smokers as Measured by Fagerstrom Test of Nicotine Dependence (FTND) Scale at Baseline Prior to the Surgery | Baseline Prior to the Surgery
  Level of smoking dependence will be measured by FTND Scale in the participant's questionnaire. FTND is a 6-item self-report measure of nicotine dependence derived from the Fagerström Tolerance Questionnaire, which comprises yes/no options (scored from 0 to 1) and multiple-choice items (scored from 0 to 3). The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the participant's physical dependence on nicotine.
Smoking Dependence Among Smokers as Measured by FTND Scale at Month 1 Post-surgery | Month 1 post-surgery
  Level of smoking dependence will be measured by FTND Scale in the participant's questionnaire. FTND is a 6-item self-report measure of nicotine dependence derived from the Fagerström Tolerance Questionnaire, which comprises yes/no options (scored from 0 to 1) and multiple-choice items (scored from 0 to 3). The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the participant's physical dependence on nicotine.
Smoking Dependence Among Smokers as Measured by FTND Scaleat Month 3 Post-surgery | Month 3 post-surgery
  Level of smoking dependence will be measured by FTND Scale in the participant's questionnaire. FTND is a 6-item self-report measure of nicotine dependence derived from the Fagerström Tolerance Questionnaire, which comprises yes/no options (scored from 0 to 1) and multiple-choice items (scored from 0 to 3). The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the participant's physical dependence on nicotine.
Smoking Dependence Among Smokers as Measured by FTND Scaleat Month 6 Post-surgery | Month 6 post-surgery
  Level of smoking dependence will be measured by FTND Scale in the participant's questionnaire. FTND is a 6-item self-report measure of nicotine dependence derived from the Fagerström Tolerance Questionnaire, which comprises yes/no options (scored from 0 to 1) and multiple-choice items (scored from 0 to 3). The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the participant's physical dependence on nicotine.
Number of Smoking Cessation Attempts at Baseline Prior to the Surgery | Baseline prior to the surgery
  Number of smoking cessation attempts at baseline prior to the surgery will be reported.
Number of Smoking Cessation Attempts at Month 1 Post-surgery | Month 1 post-surgery
  Number of smoking cessation attempts at Month 1 post-surgery will be reported.
Number of Smoking Cessation Attempts at Month 3 Post-surgery | Month 3 post-surgery
  Number of smoking cessation attempts at Month 3 post-surgery will be reported.
Number of Smoking Cessation Attempts at Month 6 Post-surgery | Month 6 post-surgery
  Number of smoking cessation attempts at Month 6 post-surgery will be reported.
Number of Participants who Used Methods and Medications for Smoking Cessation at Baseline | Baseline
  Number of participants who used prior methods and medications for smoking cessation at baseline will be reported.
Number of Participants who Used Current Methods and Medications for Smoking Cessation at Month 1 Post-surgery | Month 1 post-surgery
  Number of participants who used current methods or medication for smoking cessation at Month 1 post-surgery will be reported.
Number of Participants who Used Current Methods and Medications for Smoking Cessation at Month 3 Post-surgery | Month 3 post-surgery
  Number of participants who used current methods or medication for smoking cessation at Month 3 post-surgery will be reported.
Number of Participants who Used Prior Methods and Medications for Smoking Cessation at Month 6 Post-surgery | Month 6 post-surgery
  Number of participants who used current methods or medication for smoking cessation at Month 6 post-surgery will be reported.
Percentage of Participants Using Nicotine Replacement Therapy (NRTs) at Baseline Prior to Surgery | Baseline prior to surgery
  Percentage of participants using NRTs, types of NRTs used and perceived effectiveness, at baseline prior to surgery will be reported.
Percentage of Participants Using NRTs at Month 1 Post-surgery | Month 1 post-surgery
  Percentage of participants using NRTs, types of NRTs used and perceived effectiveness, at Month 1 post surgery will be reported.
Percentage of Participants Using NRTs at Month 3 Post-surgery | Month 3 post-surgery
  Percentage of participants using NRTs, types of NRTs used and perceived effectiveness, at Month 3 post surgery will be reported.
Percentage of Participants Using NRTs, Types of NRTs Used and Perceived Effectiveness at Month 6 Post-surgery | Month 6 post-surgery
  Percentage of participants using NRTs, types of NRTs used and perceived effectiveness, at Month 6 post surgery will be reported.
Percentage of Participants with Self-reported Smoking Abstinence and Point Prevalence at Month 1 Post-surgery | Month 1 post-surgery
  Percentage of participants with self-reported smoking abstinence and 7-days/30-day point prevalence of smoking at Month 1 post-surgery will be reported.
Percentage of Participants with Self-reported Smoking Abstinence and Point Prevalence at Month 3 Post-surgery | Month 3 post-surgery
  Percentage of participants with self-reported smoking abstinence and point prevalence of smoking at Month 3 post-surgery will be reported.
Percentage of Participants with Self-reported Smoking Abstinence and Point Prevalence at Month 6 Post-surgery | Month 6 post-surgery
  Percentage of participants with self-reported smoking abstinence and point prevalence of smoking at Month 6 post-surgery will be reported.
Percentage of Participants with Smoking Relapse at Month 1 Post-surgery | Month 1 post-surgery
  Percentage of participants with smoking relapse at Month 1 post-surgery will be reported.
Percentage of Participants with Smoking Relapse at Month 3 Post-surgery | Month 3 post-surgery
  Percentage of participants with smoking relapse at Month 3 post-surgery will be reported.
Percentage of Participants with Smoking Relapse at Month 6 Post-surgery | Month 6 post-surgery
  Percentage of participants with smoking relapse at Month 6 post-surgery will be reported.
Overall Incidence of Postoperative Complications (PCs) and Postoperative Pulmonary Complications (PPCs) Post-surgery (at 1 Day Prior to Discharge)and by Baseline Smoking Status | At 1 day prior to discharge
  Overall incidence of PCs and PPCs post-surgery (at 1 day prior to discharge) and by baseline smoking status will be reported.
Overall Incidence of PCs and PPCs Post-surgery (Within 2 Weeks After Surgery) and by Baseline Smoking Status | Within 2 weeks after surgery
  Overall incidence of PCs and PPCs post-surgery (within 2 weeks after surgery) and by baseline smoking status will be reported.
Overall Incidence of PCs and PPCs Post-surgery (Within 1 Month Post-surgery) and by Baseline Smoking Status | Within 1 month post-surgery
  Overall incidence of PCs and PPCs post-surgery (within 1 month post-surgery) and by baseline smoking status will be reported.
Overall Incidence of PCs and PPCs Post-surgery (Within 3 Months Post-surgery) and by Baseline Smoking Status | Within 3 months post-surgery
  Overall incidence of PCs and PPCs post-surgery (within 3 months post-surgery) and by baseline smoking status will be reported.
Overall Incidence of PCs and PPCs Post-surgery (Within 6 Months Post-surgery) and by Baseline Smoking Status | Within 6 months post-surgery
  Overall incidence of PCs and PPCs post-surgery (within 6 months post-surgery) and by baseline smoking status will be reported.
Percentage of Participants who Received Advice from HCPs to Quit Smoking at Baseline Prior to Surgery | Baseline prior to surgery
  Percentage of participants who received advice from HCPs to quit smoking at baseline prior to surgery will be reported.
Percentage of Participants who Received Advice from HCPs to Quit Smoking at Month 1 Post-surgery | Month 1 post-surgery
  Percentage of participants who received advice from HCPs to quit smoking at Month 1 post-surgery will be reported.
Percentage of Participants who Received Advice from HCPs to Quit Smoking at Month 3 post-surgery | Month 3 post-surgery
  Percentage of participants who received advice from HCPs to quit smoking at Month 3 post-surgery will be reported.
Percentage of Participants who Received Advice from HCPs to Quit Smoking at Month 6 post-surgery | Month 6 post-surgery
  Percentage of participants who received advice from HCPs to quit smoking at Month 6 post-surgery will be reported.
Percentage of Specific Smoking Cessation Methods and Service Participants Received from HCPs at Baseline Prior to Surgery | Baseline prior to surgery
  Percentage of specific smoking cessation methods and service participants received from HCPs at baseline prior to surgery will be reported.
Percentage of Specific Smoking Cessation Methods and Service Participants Received from HCPs at Baseline Prior to Surgery | Month 1 post-surgery
  Percentage of specific smoking cessation methods and service participants received from HCPs at Month 1 post-surgery will be reported.
Percentage of Specific Smoking Cessation Methods and Service Participants Received from HCPs at Month 3 post-surgery | Month 3 post-surgery
  Percentage of specific smoking cessation methods and service participants received from HCPs at Month 3 post-surgery will be reported.
Percentage of Specific Smoking Cessation Methods and Service Participants Received from HCPs at Month 6 post-surgery | Month 6 post-surgery
  Percentage of specific smoking cessation methods and service participants received from HCPs at Month 6 post-surgery will be reported.
Percentage of Participant's Satisfaction on the Smoking Cessation Methods Received from HCPs at Baseline Prior to Surgery | Baseline prior to surgery
  Percentage of participant's satisfaction on the smoking cessation methods received from HCPs at baseline prior to surgery will be reported.
Percentage of Participant's Satisfaction on the Smoking Cessation Methods Received from HCPs at Month 1 Post-surgery | Month 1 post-surgery
  Percentage of participant's satisfaction on the smoking cessation methods received from HCPs at Month 1 post-surgery will be reported.
Percentage of Participant's Satisfaction on the Smoking Cessation Methods Received from HCPs at Month 3 Post-surgery | Month 3 post-surgery
  Percentage of participant's satisfaction on the smoking cessation methods received from HCPs at Month 3 post-surgery will be reported.
Percentage of Participant's Satisfaction on the Smoking Cessation Methods Received from HCPs at Month 6 Post-surgery | Month 6 post-surgery
  Percentage of participant's satisfaction on the smoking cessation methods received from HCPs at Month 6 post-surgery will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson (China) Investment Ltd. Clinical Trial, Study Director — Johnson & Johnson (China) Investment Ltd.
Locations (3):
- China (3):
  - Xuanwu Hospital ,Capital Medical University, Beijing
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai

IPD SHARING:
Plan to Share IPD: No